CLINICAL TRIAL: NCT06422819
Title: Probing the Heart Rate Variability Biofeedback as an Innovative and Non-invasive Treatment for Functional Neurological Disorders Guided by a Multimodal Approach of Autonomic Nervous System.
Brief Title: Clinical Evaluation of HRV Biofeedback in Functional Neurological Disorders Compared to Placebo
Acronym: HRV_BFB_FND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-12156
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Functional Neurological Disorder
Keywords: Functional Neurological Disorder; Emotional dysregulation; Autonomic nervous system; Endophenotypes; Biofeedback of Heart Rate Variability; Transdiagnostic approach
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Intervention Model Description: This study consists of 5 visits (V1, V2, V3, V4, V5). At V1, participants will be randomized into two groups: HRV-BFB (experimental group) or Pseudo HRV-BFB (control group). Participants will remain single-blinded after randomization. Depending on the assigned group, participants will practice one specific intervention during the first 30-day period (V1-V2). At V2, participants will switch to the other arm and practice the second intervention during the second 30-day period (V2-V3). At V3, both interventions will end, and participants will be unblinded and encouraged to continue HRV-BFB at home. Clinical evaluation will be repeated 5 times at day 1 (V1), days 30 +/- 10 (V2), days 60 +/- 10 (V2), 6 months (V4) and 1 year (V5). The research team will exercise extreme caution to ensure consistent instructions and feedback, minimizing biases associated with lack of double-blinding.
Who Masked: Participant
Masking Description: The participants won't be informed of the condition to which they belong. A debriefing will be done at the end of the last intervention (V3) for each participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (HRV-BFB training) (Experimental): Participants assigned to the experimental group will undergo HRV Biofeedback training using the Inner Balance Coherence Plus® software. This software incorporates a Bluetooth plethysmograph ear sensor, which will transmit cardiac pulse data to the Inner Balance Coherence Plus smartphone app, where the EmWave Pro® Plus software will extract HRV in real-time. This software will display the participant's HRV-BFB curve on their smartphone. The installation of the program and necessary instructions for its use will be provided at the first visit (V1). Fractional training sessions of 8 minutes will be recommended, twice daily for 30 days (during the period V1-V2 or the period V2-V3). Respiratory instructions will differ between the two interventions. During the HRV-BFB intervention, participants will be instructed to maximize their HRV.
  Interventions: Other: Heart rate variability Biofeedback [HRV-BFB]
- Placebo Control group (Pseudo HRV-BFB training) (Placebo Comparator): Participants assigned to the placebo group will undergo a pseudo HRV Biofeedback training using the same Inner Balance Coherence Plus® software and ear sensor. The software will similarly display the participant's HRV-BFB curve on their smartphone. The installation of the program and necessary instructions for its use will be provided at the first visit (V1). To manage placebo effects, the same fractional training sessions of 8 minutes will be recommended, twice daily for 30 days (during the period V1-V2 or the period V2-V3). Respiratory instructions will differ between the two interventions. During the placebo pseudo BFB training, participants will be instructed to no have specific effect on HRV.
  Interventions: Other: Pseudo HRV-BFB

INTERVENTIONS:
Other: Heart rate variability Biofeedback [HRV-BFB] — Biofeedback (BFB), sometimes referred to as "biological feedback technique," is a non-invasive and non-pharmacological approach based on physiological recordings that provide real-time feedback enabling people to learn how to control their physiological processes, which are typically unconscious and beyond their control. HRV-BFB specifically targets heart rate variability (HRV), which can help regulate the autonomic nervous system (including vagal tone and sympathetic-parasympathetic balance) as well as emotional states. HRV-BFB has been clinically and experimentally validated as a physiological intervention and has demonstrated its effectiveness. However, it has never been studied in an adult FND population.
  Arms: Experimental group (HRV-BFB training)
Other: Pseudo HRV-BFB — The pseudo HRV-BFB intervention aims to implement the same HRV BFB methods with no specific effect on HRV.
  Arms: Placebo Control group (Pseudo HRV-BFB training)

SUMMARY:
Evaluation of the clinical effects of the Heart Rate Variability biofeedback training with patients suffering from Functional neurological Disorders compared with placebo.

DETAILED DESCRIPTION:
Although Functional Neurological Disorders (FND) represent one of the most common reasons for consultation in Neurology, the pathological mechanisms remain unexplained. Recent studies suggest disrupted emotional processes in patients with FND and disturbed autonomic nervous system profiles, highligting the hypothesis of autonomic endophenotypes among the FND population.

The Heart Rate Variability Biofeedback (HRV-BFB) is an innovative and non-invasive approach, based on the self-regulation of autonomic physiological processes. It has shown promising results in clinical and non-clinical populations but has never been assessed in an adult FND population.

Therefore, this approach appears particularly promising for understanding the mechanisms underlying FND and developing personalized therapy.

The main objective is to investigate the clinical effects of HRV-BFB on FND patients compared to placebo in a single-blind crossover design.

The investigators predict that depending on their autonomic profile, patients will respond to HRV-BFB to varying degrees.

Firstly, patients with FND will prospectively undergo an comprehensive clinical evaluation considering symptoms, functional capacity, quality of life, and an assessment of the physical and psychological comorbidities. Then patients will complete an emotional task and undergo multimodal autonomic measures. Cluster analyses will be conducted to identify both dysfunctional and functional autonomic profiles associated with the clinical exploration, enabling confirmation of the endophenotypes hypothesis and allowing for specific characterization of the profils. The clinical evaluation of the beneficial effects of HRV BFB will rely on repeated mesures of symptoms, functional capacity, and quality of life at scheduled points in time before and after the both interventions (HRV-BFB and pseudo-BFB). The emotional task and autonomic measures will be repeated simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Functional Neurological Disorders (FND) diagnosis must be medically established
* Participants must have a smartphone (android ou Iphone)
* Participants must be of the age of majority
* Participants must have signed an informed consent
* Sufficiently fluent in French to understand study documents and instructions
* Consistency in performing repeated questionnaires
* Normal or corrected-to-normal visual acuity

Exclusion Criteria:

* Specially protected participants: juveniles, pregnant womens, nursing mothers, law's protection peoples
* Participants suffering from a severe psychiatric disease needing specialised attention
* History of severe neurosurgical pathology
* Alcohol dependence or drug use
* Participants suffering from or have suffered from a severe disease causing autonomic dysfunctions (heart failure, asthma, blood disease, renal failure, peripheral neuropathy, vagotomy, thyroid disorder, alcoholism, liver disease, amyloidosis)
* Participants taking medication which could be impact autonomic nervous system activity (anticholinergic, antiarrhythmics, clonidine, beta-blockers, tricyclic anti-depressants, metronidazole)
* Participants placing under judicial or administrative supervisions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Patient Clinical Global Impression Score | Day 1 (V1)
  The impression improvement and severity of the core symptoms will be measured by the participant using the Clinical Global Impression Improvement and/or Severity scale (CGI-I & CGI-S; French version Busner & Targum, 2007). This scale includes 2 items.
Patient Clinical Global Impression Score | Up to 40 days from V1 (V2)
  The impression improvement and severity of the core symptoms will be measured by the participant using the Clinical Global Impression Improvement and/or Severity scale ( (CGI-I & CGI-S; French version Busner & Targum, 2007). This scale includes 2 items.
Patient Clinical Global Impression Score | Up to 80 days from V1 (V3)
  The impression improvement and severity of the core symptoms will be measured by the participant using the Clinical Global Impression Improvement and/or Severity scale ( (CGI-I & CGI-S; French version Busner & Targum, 2007). This scale includes 2 items.
Patient Clinical Global Impression Score | Up to 180 days from V1 (V4)
  The impression improvement and severity of the core symptoms will be measured by the participant using the Clinical Global Impression Improvement and/or Severity scale ( (CGI-I & CGI-S; French version Busner & Targum, 2007). This scale includes 2 items.
Patient Clinical Global Impression Score | Up to 360 days from V1 (V5)
  The impression improvement and severity of the core symptoms will be measured by the participant using the Clinical Global Impression Improvement and/or Severity scale ( (CGI-I & CGI-S; French version Busner & Targum, 2007). This scale includes 2 items.
Clinician Clinical Global Impression Score | Day 1 (V1)
  The impression improvement and severity of the core symptoms will be measured by the clinician using the Clinical Global Impression Improvement and/or Severity scale (CGI; French version Busner & Targum, 2007). This scale includes 2 items.
Clinician Clinical Global Impression Score | Up to 40 days from V1 (V2)
  The impression improvement and severity of the core symptoms will be measured by the clinician using the Clinical Global Impression Improvement and/or Severity scale (CGI; French version Busner & Targum, 2007). This scale includes 2 items.
Clinician Clinical Global Impression Score | Up to 80 days from V1 (V3)
  The impression improvement and severity of the core symptoms will be measured by the clinician using the Clinical Global Impression Improvement and/or Severity scale (CGI; French version Busner & Targum, 2007). This scale includes 2 items.
Clinician Clinical Global Impression Score | Up to 180 days from V1 (V4)
  The impression improvement and severity of the core symptoms will be measured by the clinician using the Clinical Global Impression Improvement and/or Severity scale (CGI; French version Busner & Targum, 2007). This scale includes 2 items.
Clinician Clinical Global Impression Score | Up to 360 days from V1 (V5)
  The impression improvement and severity of the core symptoms will be measured by the clinician using the Clinical Global Impression Improvement and/or Severity scale (CGI; French version Busner & Targum, 2007). This scale includes 2 items.
Quality of life Score | Day 1 (V1)
  The Quality of life Score will be measured using the 36-Item Short Form Survey (SF-36; Jenkinson et al., 1993; French version Leplège et al., 1998). This scale includes 36 items.
Quality of life Score | Up to 40 days from V1 (V2)
  The Quality of life Score will be measured using the 36-Item Short Form Survey (SF-36; Jenkinson et al., 1993; French version Leplège et al., 1998). This scale includes 36 items.
Quality of life Score | Up to 80 days from V1 (V3)
  The Quality of life Score will be measured using the 36-Item Short Form Survey (SF-36; Jenkinson et al., 1993; French version Leplège et al., 1998). This scale includes 36 items.
Quality of life Score | Up to 180 days from V1 (V4)
  The Quality of life Score will be measured using the 36-Item Short Form Survey (SF-36; Jenkinson et al., 1993; French version Leplège et al., 1998). This scale includes 36 items.
Quality of life Score | Up to 360 days from V1 (V5)
  The Quality of life Score will be measured using the 36-Item Short Form Survey (SF-36; Jenkinson et al., 1993; French version Leplège et al., 1998). This scale includes 36 items.
Self-perception of Occupation Score | Day 1 (V1)
  The Self-perception of Occupation will be measured using the Occupational Self- Assessment scale (OSA; French version Baron et al.,2006). This scale includes 21 items.
Self-perception of Occupation Score | Up to 40 days from V1 (V2)
  The Self-perception of Occupation will be measured using the Occupational Self- Assessment scale (OSA; French version Baron et al.,2006). This scale includes 21 items.
Self-perception of Occupation Score | Up to 80 days from V1 (V3)
  The Self-perception of Occupation will be measured using the Occupational Self- Assessment scale (OSA; French version Baron et al.,2006). This scale includes 21 items.
Self-perception of Occupation Score | Up to 180 days from V1 (V4)
  The Self-perception of Occupation will be measured using the Occupational Self- Assessment scale (OSA; French version Baron et al.,2006). This scale includes 21 items.
Self-perception of Occupation Score | Up to 360 days from V1 (V5)
  The Self-perception of Occupation will be measured using the Occupational Self- Assessment scale (OSA; French version Baron et al.,2006). This scale includes 21 items.

SECONDARY OUTCOMES:
Other physical symptoms score | Day 1 (V1)
  The other physical symptoms will be measured using the Patient Health Questionnaire (PHQ-15; French version Kroenke et al., 2002). This scale includes 15 items.
Other physical symptoms score | Up to 40 days from V1 (V2)
  The other physical symptoms will be measured using the Patient Health Questionnaire (PHQ-15; French version Kroenke et al., 2002). This scale includes 15 items.
Other physical symptoms score | Up to 80 days from V1 (V3)
  The other physical symptoms will be measured using the Patient Health Questionnaire (PHQ-15; French version Kroenke et al., 2002). This scale includes 15 items.
Other physical symptoms score | Up to 180 days from V1 (V4)
  The other physical symptoms will be measured using the Patient Health Questionnaire (PHQ-15; French version Kroenke et al., 2002). This scale includes 15 items.
Other physical symptoms score | Up to 360 days from V1 (V5)
  The other physical symptoms will be measured using the Patient Health Questionnaire (PHQ-15; French version Kroenke et al., 2002). This scale includes 15 items.
Depressive symptoms score | Day 1 (V1)
  The Depressive symptoms score will be measured using the for Epidemiologic Studies-- Depression (CES-D; Radloff, 1977; French version Führer & Rouillon, 1989). This scale includes 20 items.
Depressive symptoms score | Up to 40 days from V1 (V2)
  The Depressive symptoms score will be measured using the for Epidemiologic Studies-- Depression (CES-D; Radloff, 1977; French version Führer & Rouillon, 1989). This scale includes 20 items.
Depressive symptoms score | Up to 80 days from V1 (V3)
  The Depressive symptoms score will be measured using the for Epidemiologic Studies-- Depression (CES-D; Radloff, 1977; French version Führer & Rouillon, 1989). This scale includes 20 items.
Depressive symptoms score | Up to 180 days from V1 (V4)
  The Depressive symptoms score will be measured using the for Epidemiologic Studies-- Depression (CES-D; Radloff, 1977; French version Führer & Rouillon, 1989). This scale includes 20 items.
Depressive symptoms score | Up to 360 days from V1 (V5)
  The Depressive symptoms score will be measured using the for Epidemiologic Studies-- Depression (CES-D; Radloff, 1977; French version Führer & Rouillon, 1989). This scale includes 20 items.
Trait anxiety score | Day 1 (V1)
  The Trait anxiety score will be measured using the Trait Anxiety Inventory (STAI- B; Spielberger, 1989; French version Bruchon-Schweitzer & Paulhan, 1993; Huyghe Lydie, 2021). This scale includes 20 items.
Trait anxiety score | Up to 40 days from V1 (V2)
  The Trait anxiety score will be measured using the Trait Anxiety Inventory (STAI- B; Spielberger, 1989; French version Bruchon-Schweitzer & Paulhan, 1993; Huyghe Lydie, 2021). This scale includes 20 items.
Trait anxiety score | Up to 80 days from V1 (V3)
  The Trait anxiety score will be measured using the Trait Anxiety Inventory (STAI- B; Spielberger, 1989; French version Bruchon-Schweitzer & Paulhan, 1993; Huyghe Lydie, 2021). This scale includes 20 items.
Trait anxiety score | Up to 180 days from V1 (V4)
  The Trait anxiety score will be measured using the Trait Anxiety Inventory (STAI- B; Spielberger, 1989; French version Bruchon-Schweitzer & Paulhan, 1993; Huyghe Lydie, 2021). This scale includes 20 items.
Trait anxiety score | Up to 360 days from V1 (V5)
  The Trait anxiety score will be measured using the Trait Anxiety Inventory (STAI- B; Spielberger, 1989; French version Bruchon-Schweitzer & Paulhan, 1993; Huyghe Lydie, 2021). This scale includes 20 items.
Quality of sleep measure | Day 1 (V1)
  The quality of sleep will be measured using the Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 2002, French versionAit-Aoudia et al., 2013). This scale includes 7 items.
Quality of sleep measure | Up to 40 days from V1 (V2)
  The quality of sleep will be measured using the Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 2002, French versionAit-Aoudia et al., 2013). This scale includes 7 items.
Quality of sleep measure | Up to 80 days from V1 (V3)
  The quality of sleep measure will be measure using the Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 2002, French versionAit-Aoudia et al., 2013). This scale includes 7 items.
Quality of sleep measure | Up to 180 days from V1 (V4)
  The quality of sleep will be measured using the Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 2002, French versionAit-Aoudia et al., 2013). This scale includes 7 items.
Quality of sleep measure | Up to 360 days from V1 (V5)
  The quality of sleep will be measured using the Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 2002, French versionAit-Aoudia et al., 2013). This scale includes 7 items.
Dissociative Experiences | Day 1 (V1)
  The Dissociative Experiences will be measured using the Dissociative Experiences Scale EDS; Steinberg et al., 1991; french version Eve Bernstein Carlson et Frank W. Putnam, 1986). This scale includes 28 items.
Dissociative Experiences | Up to 40 days from V1 (V2)
  The Dissociative Experiences will be measured using the Dissociative Experiences Scale EDS; Steinberg et al., 1991; french version Eve Bernstein Carlson et Frank W. Putnam, 1986). This scale includes 28 items.
Dissociative Experiences | Up to 80 days from V1 (V3)
  The Dissociative Experiences will be measured using the Dissociative Experiences Scale EDS; Steinberg et al., 1991; french version Eve Bernstein Carlson et Frank W. Putnam, 1986). This scale includes 28 items.
Dissociative Experiences | Up to 180 days from V1 (V4)
  The Dissociative Experiences will be measured using the Dissociative Experiences Scale EDS; Steinberg et al., 1991; french version Eve Bernstein Carlson et Frank W. Putnam, 1986). This scale includes 28 items.
Dissociative Experiences | Up to 360 days from V1 (V5)
  The Dissociative Experiences will be measured using the Dissociative Experiences Scale EDS; Steinberg et al., 1991; french version Eve Bernstein Carlson et Frank W. Putnam, 1986). This scale includes 28 items.
Alexithymia score | Day 1 (V1)
  Alexithymia score will be measured using the Toronto Alexithymia Scale (TAS-20; French version Loas, 1996). This scale includes 20 items.
Brief Illness Perception score | Day 1 (V1)
  Brief Illness Perception score will be measured using the Brief Illness Perception Questionnaire (B-IPQ) (Moss-Morris et al., 2002 ; French version Demoulin et al., 2015). This scale includes 9 items.
Brief Illness Perception score | Up to 40 days from V1 (V2)
  Brief Illness Perception score will be measured using the Brief Illness Perception Questionnaire (B-IPQ) (Moss-Morris et al., 2002 ; French version Demoulin et al., 2015). This scale includes 9 items.
Brief Illness Perception score | Up to 80 days from V1 (V3)
  Brief Illness Perception score will be measured using the Brief Illness Perception Questionnaire (B-IPQ) (Moss-Morris et al., 2002 ; French version Demoulin et al., 2015). This scale includes 9 items.
Brief Illness Perception score | Up to 180 days from V1 (V4)
  Brief Illness Perception score will be measured using the Brief Illness Perception Questionnaire (B-IPQ) (Moss-Morris et al., 2002 ; French version Demoulin et al., 2015). This scale includes 9 items.
Brief Illness Perception score | Up to 360 days from V1 (V5)
  Brief Illness Perception score will be measured using the Brief Illness Perception Questionnaire (B-IPQ) (Moss-Morris et al., 2002 ; French version Demoulin et al., 2015). This scale includes 9 items.
Emotion Regulation Profile | Day 1 (V1)
  The Emotion Regulation Profile score will be measured using the Emotion Regulation Profile-Revised (ERP-R) (French version Nelis et al., 2011). This scale includes 15 items.
Emotion Regulation Profile | Up to 40 days from V1 (V2)
  The Emotion Regulation Profile score will be measured using the Emotion Regulation Profile-Revised (ERP-R) (French version Nelis et al., 2011). This scale includes 15 items.
Emotion Regulation Profile | Up to 80 days from V1 (V3)
  The Emotion Regulation Profile score will be measured using the Emotion Regulation Profile-Revised (ERP-R) (French version Nelis et al., 2011). This scale includes 15 items.
Emotion Regulation Profile | Up to 180 days from V1 (V4)
  The Emotion Regulation Profile score will be measured using the Emotion Regulation Profile-Revised (ERP-R) (French version Nelis et al., 2011). This scale includes 15 items.
Emotion Regulation Profile | Up to 360 days from V1 (V5)
  The Emotion Regulation Profile score will be measured using the Emotion Regulation Profile-Revised (ERP-R) (French version Nelis et al., 2011). This scale includes 15 items.
Childhood Trauma profile | Day 1 (V1)
  The Childhood Trauma profile will be measured using the Childhood Trauma Questionnaire-Short Form (CTQ; Frenc version Paquette et al., 2004). This scale includes 28 items.
Positive Affect and Negative Affects | Day 1 (V1) before the emotional induction task
  The Positive Affect and Negative Affects will be measured using the Positive Affect and Negative Affect Schedule (PANAS; Watson et al., 1988. French version Caci & Bayle, 2007). To measure a global affective state, a score of positivity will be calculated by subtracting negative affect score from positive affect score. This scale includes 20 items.
Positive Affect and Negative Affects | Day 1 (V1) after the emotional induction task
  The Positive Affect and Negative Affects will be measured using the Positive Affect and Negative Affect Schedule (PANAS; Watson et al., 1988. French version Caci & Bayle, 2007). To measure a global affective state, a score of positivity will be calculated by subtracting negative affect score from positive affect score. This scale includes 20 items.
Positive Affect and Negative Affects | Up to 40 days from V1 (V2) before the emotional re-exposure task
  The Positive Affect and Negative Affects will be measured using the Positive Affect and Negative Affect Schedule (PANAS; Watson et al., 1988. French version Caci & Bayle, 2007). To measure a global affective state, a score of positivity will be calculated by subtracting negative affect score from positive affect score. This scale includes 20 items.
Positive Affect and Negative Affects | Up to 40 days from V1 (V2) after the emotional re-exposure task
  The Positive Affect and Negative Affects will be measured using the Positive Affect and Negative Affect Schedule (PANAS; Watson et al., 1988. French version Caci & Bayle, 2007). To measure a global affective state, a score of positivity will be calculated by subtracting negative affect score from positive affect score. This scale includes 20 items.
High Frequency [HF] (>0.15 Hz) | Day 1 (V1)
  High Frequency (>0.15 Hz), frequency-domain parameter. HF will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
High Frequency [HF] (>0.15 Hz) | Up to 40 days from V1 (V2)
  High Frequency (>0.15 Hz), frequency-domain parameter. HF will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
High Frequency [HF] (>0.15 Hz) | Up to 80 days from V1 (V3)
  High Frequency (>0.15 Hz), frequency-domain parameter. HF will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
High Frequency [HF] (>0.15 Hz) | Up to 180 days from V1 (V4)
  High Frequency (>0.15 Hz), frequency-domain parameter. HF will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
High Frequency [HF] (>0.15 Hz) | Up to 360 days from V1 (V5)
  High Frequency (>0.15 Hz), frequency-domain parameter. HF will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Root Mean Square of Successive Differences [RMSSD] | Day 1 (V1)
  Root Mean Square of Successive Differences, Frequency-domain parameter. RMSSD will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Root Mean Square of Successive Differences [RMSSD] | Up to 40 days from V1 (V2)
  Root Mean Square of Successive Differences, Frequency-domain parameter. RMSSD will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Root Mean Square of Successive Differences [RMSSD] | Up to 80 days from V1 (V3)
  Root Mean Square of Successive Differences, Frequency-domain parameter. RMSSD will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Root Mean Square of Successive Differences [RMSSD] | Up to 180 days from V1 (V4)
  Root Mean Square of Successive Differences, Frequency-domain parameter. RMSSD will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Root Mean Square of Successive Differences [RMSSD] | Up to 360 days from V1 (V5)
  Root Mean Square of Successive Differences, Frequency-domain parameter. RMSSD will be measured using the electrocardiogram [ECG]: ECG data will be recorded using 3 single use and adhesive electrodes placed on the inner side of the right wrist, on the right shoulder and on the left side in accordance with the DII standard position (Einthoven). Physiological data recorded are related to the heart rate variability [HRV].
Skin conductance responses [SCR] frequency | Day 1 (V1)
  Skin conductance responses [SCR] frequency : number of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] frequency | Up to 40 days from V1 (V2)
  Skin conductance responses [SCR] frequency : number of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] frequency | Up to 80 days from V1 (V3)
  Skin conductance responses [SCR] frequency : number of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] frequency | Up to 180 days from V1 (V4)
  Skin conductance responses [SCR] frequency : number of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] frequency | Up to 360 days from V1 (V5)
  Skin conductance responses [SCR] frequency : number of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] amplitude | Day 1 (V1)
  Skin conductance responses amplitude: amplitude of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] amplitude | Up to 40 days from V1 (V2)
  Skin conductance responses amplitude: amplitude of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] amplitude | Up to 80 days from V1 (V3)
  Skin conductance responses amplitude: amplitude of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] amplitude | Up to 180 days from V1 (V4)
  Skin conductance responses amplitude: amplitude of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Skin conductance responses [SCR] amplitude | Up to 360 days from V1 (V5)
  Skin conductance responses amplitude: amplitude of the spontaneous galvanic skin responses by periods. SCR will be measured using the Galvanic skin responses [GSR]: GSR data will be recorded using 2 skin sensors placed on the third phalanx of the forefinger and of the middle finger of the left hand. Physiological data recorded are related to the cholinergic sympathetic activity (tonic GSR / phasic GSR).
Delta frequency (0-4Hz) | Day 1 (V1)
  Delta frequency 0-4 Hertz band
  Delta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Delta frequency (0-4Hz) | Up to 40 days from V1 (V2)
  Delta frequency 0-4 Hertz band
  Delta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Delta frequency (0-4Hz) | Up to 80 days from V1 (V3)
  Delta frequency 0-4 Hertz band
  Delta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Theta frequency (4-7Hz) | Day 1 (V1)
  Theta frequency 4-7 Hertz band
  Theta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Theta frequency (4-7Hz) | Up to 40 days from V1 (V2)
  Theta frequency 4-7 Hertz band
  Theta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Theta frequency (4-7Hz) | Up to 80 days from V1 (V3)
  Theta frequency 4-7 Hertz band
  Theta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Alpha frequency (8-12Hz) | Day 1 (V1)
  Alpha frequency 8-12 Hertz band Alpha frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Alpha frequency (8-12Hz) | Up to 40 days from V1 (V2)
  Alpha frequency 8-12 Hertz band Alpha frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Alpha frequency (8-12Hz) | Up to 80 days from V1 (V3)
  Alpha frequency 8-12 Hertz band Alpha frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Beta frequency (13-30Hz) | Day 1 (V1)
  Beta frequency 13-30 Hertz band Beta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Beta frequency (13-30Hz) | Up to 40 days from V1 (V2)
  Beta frequency 13-30 Hertz band Beta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Beta frequency (13-30Hz) | Up to 80 days from V1 (V3)
  Beta frequency 13-30 Hertz band Beta frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Gamma frequency (>30Hz) | Day 1 (V1)
  Gamma frequency >30 Hertz band
  Gamma frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Gamma frequency (>30Hz) | Up to 40 days from V1 (V2)
  Gamma frequency >30 Hertz band
  Gamma frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.
Gamma frequency (>30Hz) | Up to 80 days from V1 (V3)
  Gamma frequency >30 Hertz band
  Gamma frequency will be measured using the electroencephalogram [EEG]: EEG data will be recorded using a EEG headsets including 128 electrodes. The EEG is related to the brain activity generated by the neural functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Dang Khoa Nguyen, Principal Investigator — Université de Montréal's affiliated hospital research centre
Locations (1):
- Université de Montréal's affiliated Hospital Research Centre (CRCHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Result] Lehrer P, Kaur K, Sharma A, Shah K, Huseby R, Bhavsar J, Sgobba P, Zhang Y. Heart Rate Variability Biofeedback Improves Emotional and Physical Health and Performance: A Systematic Review and Meta Analysis. Appl Psychophysiol Biofeedback. 2020 Sep;45(3):109-129. doi: 10.1007/s10484-020-09466-z. PMID 32385728
- [Result] Laborde S, Mosley E, Thayer JF. Heart Rate Variability and Cardiac Vagal Tone in Psychophysiological Research - Recommendations for Experiment Planning, Data Analysis, and Data Reporting. Front Psychol. 2017 Feb 20;8:213. doi: 10.3389/fpsyg.2017.00213. eCollection 2017. PMID 28265249
- [Result] Pick S, Anderson DG, Asadi-Pooya AA, Aybek S, Baslet G, Bloem BR, Bradley-Westguard A, Brown RJ, Carson AJ, Chalder T, Damianova M, David AS, Edwards MJ, Epstein SA, Espay AJ, Garcin B, Goldstein LH, Hallett M, Jankovic J, Joyce EM, Kanaan RA, Keynejad RC, Kozlowska K, LaFaver K, LaFrance WC Jr, Lang AE, Lehn A, Lidstone S, Maurer CW, Mildon B, Morgante F, Myers L, Nicholson C, Nielsen G, Perez DL, Popkirov S, Reuber M, Rommelfanger KS, Schwingenshuh P, Serranova T, Shotbolt P, Stebbins GT, Stone J, Tijssen MA, Tinazzi M, Nicholson TR. Outcome measurement in functional neurological disorder: a systematic review and recommendations. J Neurol Neurosurg Psychiatry. 2020 Jun;91(6):638-649. doi: 10.1136/jnnp-2019-322180. Epub 2020 Feb 28. PMID 32111637
- [Result] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Steinberg M, Rounsaville B, Cicchetti D. Detection of dissociative disorders in psychiatric patients by a screening instrument and a structured diagnostic interview. Am J Psychiatry. 1991 Aug;148(8):1050-4. doi: 10.1176/ajp.148.8.1050. PMID 1853955
- [Result] Loas G, Otmani O, Verrier A, Fremaux D, Marchand MP. Factor analysis of the French version of the 20-Item Toronto Alexithymia Scale (TAS-20). Psychopathology. 1996;29(2):139-44. doi: 10.1159/000284983. PMID 8861519
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Boucsein W, Fowles DC, Grimnes S, Ben-Shakhar G, roth WT, Dawson ME, Filion DL; Society for Psychophysiological Research Ad Hoc Committee on Electrodermal Measures. Publication recommendations for electrodermal measurements. Psychophysiology. 2012 Aug;49(8):1017-34. doi: 10.1111/j.1469-8986.2012.01384.x. Epub 2012 Jun 8. PMID 22680988
- [Result] American Clinical Neurophysiology Society. Guideline 6: A proposal for standard montages to be used in clinical EEG. J Clin Neurophysiol. 2006 Apr;23(2):111-7. doi: 10.1097/00004691-200604000-00007. No abstract available. PMID 16612227
- See also: Radloff LS. The CES-D scale: a self report depression scale for research in the general population. App Psycho Meas 1977;1:384-401. — http://conservancy.umn.edu/handle/11299/98561
- See also: Paul Lehrer. Protocol for Heart Rate Variability Biofeedback Training. DOI:10.5298/1081-5937-41.3.08 — http://www.researchgate.net/publication/289937389_Protocol_for_Heart_Rate_Variability_Biofeedback_Training
- See also: Alain Leplège 2001. Le questionnaire MOS SF-36, manuel d'utilisation et guide d'interprétation des scores — http://www.researchgate.net/publication/281433197_Le_questionnaire_MOS_SF-36_manuel_d'utilisation_et_guide_d'interpretation_des_scores_French
- See also: Kathi Baron 2006 A User's Manual for the Occupational Self Assessment (OSA) : (Version 2.2) — http://search.worldcat.org/fr/title/A-User%27s-Manual-for-the-Occupational-Self-Assessment-(OSA)-:-(Version-2.2)/oclc/475547618
- See also: C Demoulin 2017. Traduction en français du " Brief Illness Perceived Questionnaire " adapté aux patients lombalgiques et étude de ses qualités métrologiques. Doi : 10.1016/S1169-8330(16)30511-7 — http://www.em-consulte.com/article/1100188/traduction-en-francais-du-%C2%A0brief-illness-perceived
- See also: Daniel Paquette 2004. Validation de la version française du CTQ et prévalence de l'histoire de maltraitance. DOI: 10.7202/008831ar — http://www.erudit.org/fr/revues/smq/2004-v29-n1-smq755/008831ar/